CLINICAL TRIAL: NCT03199859
Title: Early Diagnosis and Treatment Standardization of Delirium
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bong-Jin Hahm, Professor, Seoul National University Hospital
Other Study IDs: 072016105
Record Dates: First submitted 2017-06-22; First posted 2017-06-27 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Delirium
Keywords: gastric cancer; postoperative; subsyndromal delirium; quality of life
MeSH Terms: conditions — Delirium; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Observe the characteristics of delirium patients, searching for early diagnostic methods or finding risk factors
2. Design a guideline for delirium, diagnosis or treatment

DETAILED DESCRIPTION:
The study is consisted of two parts; First, observational study of gastric cancer patients admitted to hospital, diagnosing the presence of delirium or subsyndromal delirium and collecting patient data, including assessment, self-report surveys, and electronic medical records.

Second, Designing a guideline for treating delirium patients in Korea using the study data and reviewing other studies, guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Curable malignant gastric cancer

Exclusion Criteria:

* Gastrointestinal stromal tumor
* Uncurable cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the gastric cancer department of general surgery at Seoul National University Hospital due for surgical resection were included.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-05-17 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Delirium Rating Scale-98 | Till 1 year after surgery
  Delirium rating tool, score of 8 for subsyndromal delirium, 15 for delirium

SECONDARY OUTCOMES:
Functional assessment of cancer therapy - gastric cancer | Till 1 year after surgery
  Quality of life measuring tool for gastric cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No